CLINICAL TRIAL: NCT01135524
Title: A Randomized, Double-blind, Multicenter, Active Comparator Study to Determine the Efficacy and Safety of BTDS 20 or OxyIR® Versus BTDS 5 in Subjects With Moderate to Severe Osteoarthritis (OA) Pain: A 52-Week Extension Phase
Brief Title: Safety of Buprenorphine Transdermal Patch (BTDS) in Osteoarthritis Pain: a 52-Week Extension Phase
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was terminated early for administrative reasons.
Sponsor: Purdue Pharma LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BUP3019S
Record Dates: First submitted 2010-06-01; First posted 2010-06-02 (Estimated); Results first posted 2010-09-23 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Opioid; Transdermal
MeSH Terms: conditions — Osteoarthritis | interventions — Buprenorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BTDS (Experimental): Buprenorphine transdermal patch
  Interventions: Drug: Buprenorphine transdermal patch

INTERVENTIONS:
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 5 mcg/h applied transdermally for 7-day wear.
  Other Names: Butrans™
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 10 mcg/h applied transdermally for 7-day wear.
  Other Names: Butrans™
Drug: Buprenorphine transdermal patch — Buprenorphine transdermal patch 20 mcg/h applied transdermally for 7-day wear.
  Other Names: Butrans™

SUMMARY:
The purpose of this phase is to evaluate the long-term safety and tolerability of BTDS. Qualified subjects are started on BTDS 5 and the dose may be titrated, if necessary, to a maximum of BTDS 20 to achieve stable pain control.

DETAILED DESCRIPTION:
Buprenorphine is a synthetic opioid analgesic with over 25 years of international clinical experience indicating it to be safe and effective in a variety of therapeutic situations for the relief of moderate to severe pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed all visits of the double-blind phase on study drug and subjects who discontinued study drug due to lack of therapeutic effect in the double-blind phase but completed all visits of the double-blind phase off study drug are eligible to enroll in the extension phase.

Exclusion Criteria:

* Subjects who prematurely discontinue study drug in the double-blind phase due to adverse event, subject's choice, administrative reason or lost to follow-up are NOT eligible to enter the extension phase
* Subjects with electrocardiograms (ECGs) that show any QT data corrected for heart rate using Fridericia formula (QTcF) interval ≥ 500 millisecond (msec) will be discontinued from the extension phase.
* Subjects requiring long-acting opioid analgesics (once- or twice-daily dosing with an every (q) 24 hour (h) or q12h drug) or transdermal fentanyl during the extension phase should be discontinued from the study.

Refer to core study for additional inclusion/exclusion information.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2004-04; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (84):
- United States (84):
  - Alabama Neurology and Pain Medicine, Alabaster, Alabama
  - Research Facility, Birmingham, Alabama
  - The Birmingham Pain Center, Birmingham, Alabama
  - University of Alabama Hospital, Birmingham, Alabama
  - HealthSouth Metro West Hospital, Fairfield, Alabama
  - Research Facility, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Research Facility, Tucson, Arizona
  - Hot Springs Pain Clinic, Hot Springs, Arkansas
  - Research Facility, Buena Park, California
  - Research Facility, Chula Vista, California
  - Research Facility, Fresno, California
  - Research Facility, Los Gatos, California
  - Research Facility, Roseville, California
  - NTOUCH Research Corporation, San Diego, California
  - Research Facility, San Diego, California
  - Research Facility, Torrence, California
  - Research Facility, Upland, California
  - Research Facility, Pueblo, Colorado
  - Research Facility, Bridgeport, Connecticut
  - Research Facility, Coral Gables, Florida
  - Research Facility, Daytona Beach, Florida
  - Research Facility, Hialeah, Florida
  - Research Facility, Jupiter, Florida
  - Research Facility, Largo, Florida
  - Research Facility, Miami, Florida
  - Research Facility, North Miami Beach, Florida
  - Research Facility, Ocala, Florida
  - Research Facility, Ormond Beach, Florida
  - Research Facility, Palm Harbor, Florida
  - Research Facility, Pembroke Pines, Florida
  - Radiant Research, Pinellas Park, Florida
  - Research Facility, Plantation, Florida
  - Research Facility, Port Orange, Florida
  - Research Facility, Tampa, Florida
  - Research Facility, West Palm Beach, Florida
  - Research Facility, Marietta, Georgia
  - Research Facility, Boise, Idaho
  - Idaho Arthritis Osteoporosis, Meridian, Idaho
  - Research Facility, Chicago, Illinois
  - Research Facility, Springfield, Illinois
  - Integrated Clinical Trials, West Des Moines, Iowa
  - Louisville Endocrinology PSC, Louisville, Kentucky
  - Research Facility, Madisonville, Kentucky
  - Research Facility, New Orleans, Louisiana
  - Dolby Providers, New Orleans, Louisiana
  - Research Facility, Baltimore, Maryland
  - Patuxent Medical Group, Columbia, Maryland
  - Research Facility, Hagerstown, Maryland
  - Research Facility, Brockton, Massachusetts
  - Crystal Lake Health Center, Benzonia, Michigan
  - Rheumatology PC, Kalamazoo, Michigan
  - Research Facility, Lansing, Michigan
  - KC Pain Centers East, Independence, Missouri
  - Research Facility, St Louis, Missouri
  - HealthCare Research LLC, St Louis, Missouri
  - Research Facility, Las Vegas, Nevada
  - Research Facility, New York, New York
  - Research Facility, Syracuse, New York
  - The Arthritis Clinic and Carolina Bone and Joint, Charlotte, North Carolina
  - Triangle Orthopaedic Associates, Durham, North Carolina
  - Research Facility, Greensboro, North Carolina
  - Research Facility, Hickory, North Carolina
  - Cornerstone Research Care, High Point, North Carolina
  - Research Facility, Cincinnati, Ohio
  - Research Facility, Columbus, Ohio
  - Research Facility, Oklahoma City, Oklahoma
  - Research Facility, Eugene, Oregon
  - Research Facility, Altoona, Pennsylvania
  - Research Facility, Duncansville, Pennsylvania
  - The Clinical Trial Center, Jenkintown, Pennsylvania
  - Research Facility, Mechanicsburg, Pennsylvania
  - New England Center for Clinical Research, Cranston, Rhode Island
  - Radiant Research, Greer, South Carolina
  - Allergy ARTS, Amarillo, Texas
  - Research Facility, Conroe, Texas
  - Family Practice Associates, Corpus Christi, Texas
  - Research Facility, Dallas, Texas
  - Research Facility, Houston, Texas
  - KRK Medical Research, Richardson, Texas
  - Research Facility, San Antonio, Texas
  - Research Facility, Spokane, Washington
  - Research Facility, Milwaukee, Wisconsin
  - Research Facility, New Berlin, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 02-Apr-2004 (first subject first visit, core study) to 05-Aug-2005 (last subject last visit, extension phase), in 82 sites in the US; 59 sites randomized at least 1 subject.
Pre-assignment Details: Subjects with moderate to severe osteoarthritis (OA) pain who required opioid analgesia; completed all visits of the double-blind phase on study drug, or who discontinued study drug due to lack of therapeutic effect in the double-blind phase and completed all visits of the double-blind phase off study drug were eligible for the extension phase.
Groups:
- Extension Phase: Open-label buprenorphine transdermal patch 5, 10, 20 mcg/h applied for 7-day wear
Period: Overall Study
Arm/Group | Extension Phase
Started | 196
Completed | 0
Not Completed | 196
Not completed — Withdrawal by Subject | 14
Not completed — Adverse Event | 20
Not completed — Lost to Follow-up | 3
Not completed — Administrative | 151
Not completed — Lack of Efficacy | 8

BASELINE CHARACTERISTICS:
Arm/Group | Extension Phase
Number analyzed (Participants) | 196
Age Continuous [Mean (Standard Deviation); unit: years] | 58.4 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 46

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Description: Safety was assessed using reports of adverse events, clinical laboratory results, findings from physical examinations, and vital sign measurements.
Time Frame: 52 weeks
Population: The Extension Safety Population (N = 196) consisted of all subjects who received at least 1 dose of the open-label BTDS extension study drug, and had at least 1 safety assessment during the extension phase.
Measure: Number; unit: participants
Arm/Group | Extension Phase
Number analyzed (Participants) | 196
participants
  Deaths | 1
  Serious Adverse Events | 14
  Other Adverse Events in ≥ 4.5% of subjects | 93

ADVERSE EVENTS:
Time Frame: Extension phase: AEs occurring after the application of the first patch during the extension phase were recorded up to 7 days after the last visit; serious AEs up to 30 days following the last study visit were followed until the event resolved.
Description: AEs were obtained through spontaneous reports and subject interview.
Arm/Group | Extension Phase
Serious Adverse Events (participants affected / at risk) | 14/196
Other Adverse Events (participants affected / at risk) | 93/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Extension Phase (N=196)
Aggravated osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Systematic and nonsystematic assessments
Atypical chest pain (General disorders) | 1 (1) — Systematic and nonsystematic assessments.
Cerebrovascular accident (Nervous system disorders) | 1 (1) — Systematic and nonsystematic assessments.
Chest pain (General disorders) | 1 (1) — Systematic and nonsystematic assessments.
Gangrene right foot (Vascular disorders) | 1 (1) — Systematic and nonsystematic assessments.
Gastroenteritis (Gastrointestinal disorders) | 1 (1) — Systematic and nonsystematic assessments.
Herniated lumbar disc (Musculoskeletal and connective tissue disorders) | 1 (1) — Systematic and nonsystematic assessments.
Left lung pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Systematic and nonsystematic assessments
Mild myocardial infarction (Cardiac disorders) | 1 (1) — Systematic and nonsystematic assessments.
Myocardial infarction (Cardiac disorders) | 1 (1) — Systematic and nonsystematic assessments.
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) — DEATH Systematic and nonsystematic assessments.
Rectal polyp (Gastrointestinal disorders) | 1 (1) — Systematic and nonsystematic assessments.
Unstable angina (Cardiac disorders) | 1 (1) — Systematic and nonsystematic assessments.
Weight loss (Investigations) | 1 (1) — Systematic and nonsystematic assessments.
Withdrawal symptoms (General disorders) | 1 (1) — Systematic and nonsystematic assessments.
Worsening hiatal hernia (Gastrointestinal disorders) | 1 (1) — Systematic and nonsystematic assessments
Worsening left hip OA (Musculoskeletal and connective tissue disorders) | 1 (1) — Systematic and nonsystematic assessments.
Worsening of lumbar stenosis (Nervous system disorders) | 1 (1) — Systematic and nonsystematic assessments.
OTHER ADVERSE EVENTS (reported when occurring in more than 4.50% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Extension Phase (N=196)
Application site erythema (General disorders) | 11 — Systematic and nonsystematic assessments.
Application site pruritus (General disorders) | 22 — Systematic and nonsystematic assessments.
Application site rash (General disorders) | 20 — Systematic and nonsystematic assessments.
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 — Systematic and nonsystematic assessments.
Constipation (Gastrointestinal disorders) | 9 — Systematic and nonsystematic assessments.
Headache (Nervous system disorders) | 31 — Systematic and nonsystematic assessments.
Joint swelling (Musculoskeletal and connective tissue disorders) | 9 — Systematic and nonsystematic assessments.
Nausea (Gastrointestinal disorders) | 12 — Systematic and nonsystematic assessments.
Pain NOS (General disorders) | 10 — Systematic and nonsystematic assessments.
Pain in limb (Musculoskeletal and connective tissue disorders) | 10 — Systematic and nonsystematic assessments.
Urinary tract infection NOS (Infections and infestations) | 10 — Systematic and nonsystematic assessments.

LIMITATIONS AND CAVEATS:
This study was terminated early for administrative reasons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days